CLINICAL TRIAL: NCT03414996
Title: The Effects of High-intensity Interval Training on Maximal Oxygen Uptake and Autonomic Nervous System in Patients With Post-acute Coronary Syndrome
Brief Title: High-intensity Interval Training in Patients With Post-acute Coronary Syndrome
Acronym: EXIT-IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MontrealHI EXIT-IV
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Acute Coronary Syndrome; Arrhythmia
Keywords: Interval training; Autonomic nervous system; Post-acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Arrhythmias, Cardiac | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental): Following 5 min warm-up at 30 % of maximal aerobic power (MAP) obtained at the cardiopulmonary exercise test, patients performed 2 sets of 10 minutes of repeated phases of 15 seconds at 100 % MAP alternating with 15 seconds of passive recovery. The 2 sets were separated by 4 min of passive recovery (no pedalling). Patients performed 5-minutes of recovery period at 30 % MAP after the second set. Total time duration was 34 minutes.
  Interventions: Other: Exercise training
- Moderate-intensity continuous exercise training (Active Comparator): Duration was adjusted to match total energy expenditure of the high-intensity interval training session. Following 5 min warm-up at 30 % of maximal aerobic power (MAP), patients performed continuous exercise at 60 % MAP during 24 minutes. Patients performed 5-minutes of recovery period at 30 % MAP after the second set. Total time duration was 34 minutes.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Patients will undergo two weekly exercise training sessions with high-intensity interval training or moderate-intensity continuous exercise training for a period of 12 weeks.

SUMMARY:
To date, no studies have evaluated the safety or efficiency (improvement of maximal oxygen uptake [VO2peak]) of a high-intensity interval training (HIIT) program in post-acute coronary syndrome (post-ACS) patients. Heart rate variability (HRV) and recovery (HRR), QT dispersion (QTd) and ventricular arrhythmias are all indices associated with an increased risk of cardiac death. HIIT has been shown to improve these risk markers and be safe in coronary heart disease patients but not yet in post-ACS patients which are considered more at risks.

The aim of this study was to compare a HIIT program to a moderate-intensity continuous exercise training (MICET) program on HRV, HRR, QTd parameters and occurrence of ventricular arrhythmias in post-ACS patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years
* Acute coronary syndrome within 6 weeks (unstable angina, or non-ST elevation myocardial infarction (NSTEMI), or ST elevation myocardial infarction (STEMI with the presence of 2/3 criteria (i.e. typical chest pain, electrocardiographic ischemic change or elevated troponin T
* Complete revascularization defined as no major epicardial coronary artery or bypass graft with a residual diameter stenosis >50% and no residual left main stenosis ≥40%
* Left ventricular ejection fraction >40%
* Stable doses of medication during the 4 weeks prior to enrolment (STEMI patients must be on a stable dose of beta-blocker)
* Able to perform a maximal cardiopulmonary exercise test, 7) capacity and willingness to sign informed consent.

Exclusion Criteria:

* Recent coronary bypass surgery (<6 months)
* Incomplete revascularisation, left ventricular ejection fraction <40%
* Significant valvular disease (mitral stenosis, moderate to severe mitral insufficiency, aortic stenosis, or aortic insufficiency)
* Uncontrolled hypertension (systolic blood pressure/diastolic blood pressure >180/110 mmHg)
* Significant resting electrocardiogram abnormalities (left bundle branch block, non-specific intraventricular conduction delay, left ventricular hypertrophy, resting ST-segment depression)
* Chronic atrial fibrillation
* Pacemaker or implantable cardioverter defibrillator
* Low functional capacity (<5 basal Metabolic Equivalent of Task [METs])
* Change of cardiac medications within 4 weeks of enrolment and any contraindication to exercise testing or exercise training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | At baseline and following 12 weeks exercise training intervention
  Change before and after exercise training

SECONDARY OUTCOMES:
Markers of autonomic nervous system | At baseline and following 12 weeks exercise training intervention
  Change before and after exercise training

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular prevention and rehabilitation center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trachsel LD, David LP, Gayda M, Boidin M, Lalonge J, Juneau M, Nigam A, Henri C. Impact of aerobic training periodisation on global and regional right ventricular strain in coronary heart disease. Appl Physiol Nutr Metab. 2021 Dec;46(12):1502-1509. doi: 10.1139/apnm-2021-0055. Epub 2021 Jul 26. PMID 34310883
- [Derived] Trachsel LD, Boidin M, Henri C, Fortier A, Lalonge J, Juneau M, Nigam A, Gayda M. Women and men with coronary heart disease respond similarly to different aerobic exercise training modalities: a pooled analysis of prospective randomized trials. Appl Physiol Nutr Metab. 2021 May;46(5):417-425. doi: 10.1139/apnm-2020-0650. Epub 2020 Oct 23. PMID 33096006
- [Derived] Trachsel LD, Nigam A, Fortier A, Lalonge J, Juneau M, Gayda M. Moderate-intensity continuous exercise is superior to high-intensity interval training in the proportion of VO2peak responders after ACS. Rev Esp Cardiol (Engl Ed). 2020 Sep;73(9):725-733. doi: 10.1016/j.rec.2019.09.013. Epub 2019 Dec 16. English, Spanish. PMID 31837947